CLINICAL TRIAL: NCT01355653
Title: AN OPEN LABEL STUDY TO COMPARE THE EFFECTS OF AGE AND BODY FAT ON THE SAFETY OF TWO HEAT WRAP DEVICES IN HEALTHY SUBJECTS
Brief Title: Heat Wrap Device Safety With Age and Body Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B3571002; TC-09-12 (Other: Alias Study Number)
Record Dates: First submitted 2011-04-28; First posted 2011-05-18 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Back Pain
Keywords: heat; device; safety; performance; heatwrap; elderly; overweight
MeSH Terms: conditions — Back Pain; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): thermal therapy
  Interventions: Device: thermal therapy
- Treatment B (Active Comparator): ThermaCare Lower Back/Hip heatwrap
  Interventions: Device: ThermaCare heatwrap

INTERVENTIONS:
Device: thermal therapy — heat therapy device, topical, two applications, at 0-3 hours and 4-6 hours on treatment day
  Arms: Treatment A
Device: ThermaCare heatwrap — heatwrap, topical, one time application, 8 hour duration
  Arms: Treatment B

SUMMARY:
This study is designed to compare the safety, as measured by skin findings and adverse events, of two different heat devices in elderly, overweight, and elderly and overweight subjects.

DETAILED DESCRIPTION:
Safety measurements

ELIGIBILITY:
Inclusion Criteria:

* Males or females in generally good health, and who are either 18-54 years of age with a body mass index of ≥ 30 kg/m2
* or 55-84 years of age and with a body mass index ≥ 30 kg/m2 or < 30 kg/m2
* Females who are not pregnant or breastfeeding
* Subject is medically cleared for study participation

Exclusion Criteria:

* No sensitivitiy or allergy to device components in contact with skin
* Diabetes
* Any active skin disease or tattoos at the test site that would affect participation

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05-05 (Actual); Primary Completion 2011-07-28 (Actual); Study Completion 2011-07-28 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with any thermal-related skin events (defined as elevated skin response, erythema ≥ 2.0 [moderate], or pain upon touch plus non-zero erythema) | morning after product wear through 15 days after last product application

SECONDARY OUTCOMES:
Percentage of subjects with any adverse event | during and after wear for 28 days after last wear

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3571002&StudyName=Heat%20Wrap%20Device%20Safety%20with%20Age%20and%20Body%20Fat